CLINICAL TRIAL: NCT04165421
Title: A Family Focused Nursing Intervention for Patients With Atrial Fibrillation - Effect of Group Education and Family Strength Orientated Therapeutic Conversations
Brief Title: Family Focused Intervention for Patients With Atrial Fibrillation
Acronym: AFFINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Stine Rosenstrøm, RN,MHSc,PhD-student, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H19007769
Record Dates: First submitted 2019-11-01; First posted 2019-11-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family intervention group (Experimental): The intervention starts with a two hour group session for AF-patients and family members designed by the PhD student and the project nurses based on clinical guidelines of AF-management and theory from multifamily group intervention. Project nurses who are also Nurse specialists will facilitate knowledge to patients and family members about AF and how to support self-management in their daily living. Furthermore the (Family focused nursing) FFN intervention will consist of 3 -5 Family Strength Orientated Therapeutic Conversations (FAM-SOTC) accordingly to the needs of patient and the family. The FAM-SOTC conversations will be used as health promoting conversations and a way to enhance family health and psychological resilense
  Interventions: Behavioral: Family intervention group
- Control group (No Intervention): The control group will receive conventional care and treatment according to guidelines.
  Conventional care is characterized by ad hoc management as per usual standards of clinical care (with access to routine medical care, hospital care, and pharmacotherapy).

INTERVENTIONS:
Behavioral: Family intervention group — Education and Family conversations
  Arms: Family intervention group

SUMMARY:
Atrial fibrillation (AF) is a major and rapidly growing cardiac disease characterized by irregular heart rhythm. Living with AF can lead to stress, anxiety and depression for both patients and their families with increased risk of lost working days, hospitalization, and worsening of the disease. However, family-focused nursing has shown to capture the family's feelings and this could change the negative circle into a positive circle.

The study aim is to examine how families experience living with a family member with AF and if family involvement through a family focused nursing intervention and group education can improve quality of life for AF patients.

Family unit interviews, a study with focus group interviews with family members, and a randomized fidelity study evaluating the effect of the family focused nursing intervention will provide evidence-based knowledge on how to implement family focused nursing into care of patients with AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia and it is a rising problem for patients in Western countries. AF is a costly public health problem with hospitalizations as the primary expenditure. The disease and treatment is complex and requires a high degree of patient adherence to prevent complications (stroke and major bleedings) and the burden of symptoms due to irregular heartbeat often leads to poor health related quality of life. Consequences of AF also often lead to impairment of physical functioning and mental health.

When illness is considered a family affair it is important for patients and their families to have a chance to talk about issues of hope, suffering and coping. A family will need support and solutions when successfully adjusting to having a family member with a chronic illness. Little is known about how families experience habituate life with AF, their concerns and feelings and their needs for support. FFN based on The Calgary Family Assessment model (CFAM) and the Calgary Family Intervention Model (CIFM) used as a theoretical model have been shown to be effective in family focused nursing interventions supporting patients and families in adjusting to life whit a disease. The effect of these models have never been tested in nursing interventions towards patients with AF and their families.

The aim of the study is to examine how AF- patients and families are influenced by AF and to test if involving family members in a FFN intervention with group education improves outcomes for patients with AF.

The study will consist of three sub-studies:

A phenomenological qualitative explorative study with family unit interviews, a study of focus group interviews with members of the family analyzed with content analysis, and a quantitative fidelity study (n=100/50 in standard care/50 in the intervention group) evaluating the effect of a family focused nursing intervention with improvement of quality of life living with AF as the primary outcome. Relevant statistical analyzes will be used.

The two qualitative studies will gather new knowledge about families need of support which will be used to shape the family focused intervention.

The study inclusion criteria are: Men and women > 18 years with newly diagnosed AF. Family members who participate in interviews and in the intervention program are defined by the patient: e.g. spouse, son, daughter, near friend or neighbor. Patients with heart failure will be excluded.

The intervention begins with a two hour group session for AF-patients and family members designed by the PhD student and the project nurses based on clinical guidelines of AF-management and theory from multifamily group intervention. Project nurses who are also Nurse specialists will facilitate knowledge to patients and family members about AF and how to support self-management in their daily living. Furthermore the FFN intervention will consist of 3 -5 Family Strength Orientated Therapeutic Conversations (FAM-SOTC) accordingly to the needs of patient and the family. The FAM-SOTC conversations will be used as health promoting conversations and a way to enhance family health and psychological resilense. Before the FFN intervention the two project nurses and the PhD student will be trained theoretically and practically in performing health promoting family conversations at Linné University in Sweden.

It is expected that the study will provide a new understanding and evidence based knowledge on how to incorporate a family focused intervention and education of patients with AF and their families into the AF management and care.

In the future, results from the studies can be used to design a randomized controlled trial which could determine the possibilities and limitations of a tailored health promotion intervention for patients with AF.

The study is expected to be initiated in February 2019 and it will be completed in three years.

The Danish Data Protection Agency and The Scientific Ethical Committee will be asked to what degree the study has a duty to notify the agency.

Participants in the sub-studies will receive written and oral information about the project and must give written informed consent regarding participation which they can retract at any time. All data will be treated confidentially and anonymized. All data are stored securely and locked in safe electronic files.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years old with newly diagnosed AF (< 6 months since diagnose) documented in the patient file and verified by a EKG.
* Family members must be > 18 years old and defined by the patient: e.g. spouse, son, daughter, near friend or neighbor.

Exclusion Criteria:

* Patients with chronic heart failure according to international guidelines
* Patients not cable to cooperate about the project

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life between baseline and follow-up at 6 months | baseline and after 6 months
  The Atrial Fibrillation Effect on QualiTY-of-Life (AFEQT) Questionnaire

SECONDARY OUTCOMES:
Change in anxiety and depression between baseline and follow-up at 6 months | baseline and after 6 months
  Hospital Anxiety Depression Scale (HADS) Questionnaire
Change in Family functioning between baseline and follow-up at 6 months | baseline and after 6 months
  Ice Expressive Family Functioning Questionnaire (ICE-EFFQ)
Change in Family perceived support between baseline and follow-up at 6 months | baseline and after 6 months
  Ice Family Perceived Support Questionnaire(ICE-FPSQ)
number of Hospital admissions between baseline and follow-up | At follow-up 6 month after basline
  Self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Stine Rosenstrøm, MHSc, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Amager Hvidovre Copenhagen Univerity Hospital, Copenhagen, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No